CLINICAL TRIAL: NCT00003630
Title: Phase I Study of Arsenic Trioxide
Brief Title: Arsenic Trioxide in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-046; CDR0000066713 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1479
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of arsenic trioxide in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of arsenic trioxide in adult and pediatric patients with advanced solid tumors. II. Determine the pattern of clinical adverse experience of arsenic trioxide in this patient population. III. Evaluate evidence of clinical responsiveness to this treatment regimen.

OUTLINE: This is a dose escalation, open label study. Patients are stratified by age (pediatric vs adult). Patients receive arsenic trioxide IV over 1-2 hours once daily for 3 consecutive days then once weekly for 5 weeks. Patients with stable or responding disease receive additional courses of therapy every 8 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more patients out of 6 experience dose limiting toxicity. Patients are followed for at least 1 month after treatment.

PROJECTED ACCRUAL: Approximately 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor Relapsed from or resistant to at least 1 course of standard anticancer therapy AND/OR Lack of standard therapy that is known to be beneficial in the underlying disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 2.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 4 months following study No active serious infections that are not controlled by antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics No concurrent radiotherapy Surgery: See Disease Characteristics Other: No other concurrent investigational agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States